CLINICAL TRIAL: NCT03969576
Title: Efficacy and Safety of Drug-eluting Bead TACE VS Conventional TACE for Unresectable Hepatocellular Carcinoma: a Multicenter, Prospective Cohort Study
Brief Title: Drug-eluting Bead Transarterial Chemoembolisation (DEB-TACE) Versus (VS) Conventional Transarterial Chemoembolisation (cTACE) for Unresectable Hepatocellualr Carcinoma (HCC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Principal Investigator, Air Force Military Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEB-TACE-HCC
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Drug-eluting bead transarterial chemoembolization; Conventional transarterial chemoembolization; Objective response
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB-TACE (Experimental): 172 subjects in this study group will be receive the treatment of drug-eluting bead TACE
  Interventions: Procedure: DEB-TACE
- cTACE (Active Comparator): 172 subjects in this study group will be receive the treatment of conventional TACE
  Interventions: Procedure: cTACE

INTERVENTIONS:
Procedure: DEB-TACE — Patients in the DEB-TACE group received a maximum dose of 4 ml of DC bead (diameter 75-500 um) loaded with a maximum dose of 150 mg of anthracyclines drugs, such as doxorubicin. The anticancer agents and the diameter of DC Bead for individual patient will be selected according to the common clinical practice of each center. Treatment endpoint consisted of stasis of flow within feeding vessel(s) or completed delivery of maximum single-session dose of 150 mg doxorubicin. TACE will be repeated "on demand" according to the radiological response.
  Other Names: drug-eluting bead transarterial chemoembolisation
  Arms: DEB-TACE
Procedure: cTACE — Patients in the cTACE group were treated with anthracyclines, such as doxorubicin, in a mixture of lipiodol. Administration of the anticancer in oil emulsion was followed by injection of embolic materials such as gelfoam or PVA particles until complete stasis in segmental or subsegmental arterial branches. the tumor-feeding vessels should be superselected whenever possible. The anticancer agents for individual patient will be selected according to the common clinical practice of each center. TACE will be repeated "on demand" according to the radiological response.
  Other Names: conventional transarterial chemoembolisation
  Arms: cTACE

SUMMARY:
this multi-center prospective cohort study is to evaluate the efficacy and the safety of drug-eluting bead TACE compared with conventional TACE in terms of objective response in unresectable HCC

ELIGIBILITY:
Inclusion Criteria:

1. Prior informed consent
2. Confirmed Diagnosis of HCC: a. Cirrhotic subjects: Clinical diagnosis by American Association for the Study of Liver Diseases (AASLD) criteria. HCC can be defined in cirrhotic subjects by one imaging technique (CT scan, MRI, or second generation contrast ultrasound) showing a nodule larger than 2 cm with contrast uptake in the arterial phase and washout in venous or late phases or two imaging techniques showing this radiological behavior for nodules of 1-2 cm in diameter. Cytohistological confirmation is required for subjects who do not fulfill these eligibility criteria. b. Non-cirrhotic subjects: For subjects without cirrhosis, histological or cytological confirmation is mandatory. Documentation of original biopsy for diagnosis is acceptable
3. Patients with unresectable Barcelona Clinic Liver Cancer (BCLC) stage A and BCLC B, and all patients have a intermediate or high tumor burden (the diameter of largest tumor plus tumor number is more than 6)
4. Child Pugh class A/B(7) class without decompensated liver cirrhosis.
5. ECOG Performance Status 0 score
6. At least one uni-dimensional lesion measurable by MRI or CT according to the RECIST 1.1 criteria
7. Male or female subject larger than 18 years of age
8. Life expectance of at least 12 weeks.
9. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial
10. Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to randomization:

    1. Hemoglobin > 9.0 g/dl
    2. Absolute neutrophil count (ANC) >1,500/mm3
    3. Platelet count≥50x109/L
    4. ALB≥28g/L
    5. Total bilirubin < 2 mg/dL
    6. Alanine aminotransferase(ALT) and aspartate aminotransferase(AST) < 5 x upper limit of normal
    7. Blood urea nitrogen(BUN) and creatinine < 1.5 x upper limit of normal
    8. International normalized ratio(INR) < 1.7, or prothrombin time（PT） < 4 seconds above control

Exclusion Criteria:

1. Portal vein or any vascular invasion
2. Presence of extra hepatic spread
3. Presence of metastasis in biliary tract or obstruction of biliary tract
4. Presence of metastasis in brain or presence of symptom of the brain metastasis but lack of further examination to exclude brain metastasis
5. Poor blood supply for the liver tumor lesions; poor blood supply refers that the tumor lesions fail to show obvious contrast uptake in the arterial phase and washout in venous or late phases by CT scan or MRI
6. Any contraindications for hepatic embolization procedures:

   1. Known hepatofugal blood flow
   2. Known porto-systemic shunt
   3. Renal failure / insufficiency requiring hemo-or peritoneal dialysis
7. History of cardiac disease:

   1. Congestive heart failure >New York Heart Association (NYHA) class 2
   2. Uncontrolled hypertension
8. Known history of HIV infection
9. Patients who have previously been receiving any treatments against HCC
10. Active clinically serious infections (> grade 2 NCI-CTCAE Version 4.0), except for hepatitis B virus (HBV) and hepatitis C virus (HCV) infection
11. Contraindication of Anthracyclines administration, such as Doxorubicin
12. Concurrent with other cancer
13. Pregnant or breast-feeding subjects
14. Women of childbearing age did not take any contraceptive measures
15. Clinically significant gastrointestinal bleeding within 12 weeks prior to start of study
16. Major surgery within 3 weeks prior to start of study drug (e.g. thoracolaparotomy is not allowed, but noninvasive surgery, e.g. biopsy, is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Tumor response will be assessed at week 4 and week 12 after initiation of treatment and thereafter every 8 weeks, up to 1 year
  the percentage of patients who achieved complete response (CR) and partial response (PR) as the best response, according to the modified Response Evaluation Criteria In Solid Tumours (mRECIST) criteria

SECONDARY OUTCOMES:
Overall survival | The last patient has been on study for 1year
  Overall survival (OS) is measured from the treatment start until all-cause death or the last follow-up date
Time to progression | The last patient has been on study for 1year
  Time to progression is measured from the treatment start to the radiologically confirmed progression
Adverse event | The adverse event will be assessed during in hospital and every 4 weeks, up to 1year
  The terms and grade of adverse event will be present according to the Common Terminology Criteria for Adverse Event (CTCAE version 4.0)
Progression-free survival | The last patient has been on study for 1year
  Progression-free survival (PFS) is measured from the treatment start until all-cause death or untreatable progression (vascular invasion, extra hepatic spread, the Eastern Cooperative Oncology Group (ECOG) performance status >2, and Child-Pugh grade over C, but except hepatic new nodule)
Time to response | The last patient has been on study for 1year
  Time to response (TTR) is measured from the treatment start to the firstly radiologically confirmed complete response or partial response.
Duration of response | The last patient has been on study for 1year
  Duration of response (DOR) is measured from the first-time confirmed complete response or partial response to the date of radiological progression

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi, China